CLINICAL TRIAL: NCT05306769
Title: Leaving Nobody Out: a Mixed-Methods Study to Inform Implementation of Diverse and Representative Recruitment to HIV Clinical Studies at a Central London Clinic
Brief Title: Leaving Nobody Out
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 298515
Record Dates: First submitted 2022-02-21; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: * HIV positive
  * ≥18 years old
  * Currently registered to receive care under Harrison Wing (and thus potential candidates for Harrison Wing clinical studies)
  * Has ≥ 1 demographic identified to be underrepresented as specified in 'trial statistics'
  * Able and willing to provide written or witnessed informed consent to participate
- Group 2: HIV positive
  * ≥18 years old
  * Currently registered to receive care under Harrison Wing
  * Currently participating in any clinical study in which Harrison Wing is the/ a participating centre1
  * Able and willing to provide written or witnessed informed consent to participate

SUMMARY:
Established recruitment methods will be used to recruit participants. The study will be non-blinded. Eligibility will be checked and consent taken by a delegated study clinician. Participants will attend a 30 minute virtual individual semi-structured interview. Additionally, all patients attending an appointment within Harrison Wing will be invited to complete an anonymous, self-administered survey on attitudes towards participation in HIV clinical studies.

DETAILED DESCRIPTION:
Study description and population to be studied:

Researchers will employ Implementation Science methodology to understand and act upon the determinants of representation in HIV clinical studies in order to improve the diversity of study recruitment at the central London clinic-embedded research unit such that it better represents the clinic population. The setting is the Harrison Wing service: a specialist outpatient service for over 3500 people living with HIV based at Guy's and St Thomas' NHS Foundation Trust. This study will evaluate the extent and characteristics of study underrepresentation in the context of our clinic; identify and engage key stakeholder communities including both patients and clinicians, and collaboratively design a strategy to facilitate uptake of diverse recruitment and diverse participation using participatory methods.

Rationale and potential benefits of this study:

The demographic characteristics of participants in HIV clinical studies do not match those of the wider population of people living with HIV (PLHIV), from clinic-level to global scales.

Women and ethnic minorities are chronically underrepresented. Those at the intersections including ethnic minority or socially excluded women have particularly low participation rates.

Underrepresentation in HIV clinical studies is well-recognized to seriously threaten clinicians' and patients' ability to make informed decisions about treatment. Sub-group analyses often lack statistical power, whereas studies that actively or exclusively target underrepresented groups can reveal critical information about HIV treatment. Evidence is accumulating of gender and ethnicity-based differences in the transmission, physiology, course of infection, efficacy and safety of treatment, access to care and long-term wellbeing for PLHIV. ViiV Healthcare recently highlighted this and called for targeted enrolment of women in clinical trials.

There is also a clear ethical imperative regarding study recruitment: clinical studies may represent a patient's best opportunity for life-saving or quality of life enhancing therapies, particularly for individuals with poor access to services.37 Equitable trial recruitment not only underpins the evidence behind equitable HIV care but often constitutes that care itself. NIHR's equality, diversity and inclusion guidance emphasizes that every eligible person should be offered equal opportunity to participate in research regardless of demographics including ethnicity, sex, socioeconomic status or sexual orientation. Underrepresentation in Covid-19 research has drawn recent attention to the importance of diverse recruitment.

Despite this clear evidence that diverse and representative HIV clinical study recruitment is critically important yet rarely achieved, implementing diverse recruitment is a complex challenge. Participants' decisions to participate in research are multidimensional, wide-ranging, culturally relevant and locally specific. Themes in considerations cited by underrepresented groups include lack of knowledge about studies, mistrust of researchers, concern for safety, altruism, and positive perceptions of medical care within studies.

Rationale for including both patients with excluded demographics and patients who participate in HIV clinical studies:

Research into potential participants' locally relevant barriers reveals important nuance and sometimes stark differences in prevailing trends in what drives study participation. For example, in some areas distrust is a dominant barrier for men and medication concerns dominant for women, yet elsewhere trust levels are similar regardless of gender.

benefits such as sociability motivate others. Stage of disease and psychological factors are important. Interventions to increase representation have been efficacious where local factors are appreciated. Interactions between patients and study providers may also be important: study providers, such as clinicians, are gatekeepers to clinical study access. Biases in referring to clinical trials disadvantages women, ethnic minorities and psychosocially complex patients providers' perceptions of patients' recruitment barriers are not always correct. Invitation to studies may be a dominant barrier to diverse recruitment. Ironically, underrepresentation exists despite under-recruited populations desiring more representative trial populations.

Justification for research methods to be used, including virtual semi-structured interviewing and self-administered surveys:

Focus groups and semi-structured interviewing have been successfully utilized in a variety of settings to identify barriers and enablers of trial recruitment through thematic analysis in underrepresented groups. These strategies are frequently combined with baseline demographic and social data, and surveys have proved a valuable resource in identifying and overcoming barriers to diverse recruitment. The Investigators have chosen a virtual format for convenience to participants and to minimise the risk of Covid-19 infection. Self-administered surveys are effective and may be preferable through enabling anonymity of participants. Such qualitative methods can successfully identify providers' biases and barriers as well as those of patients. Assessing the representativeness of HIV patients in clinical studies using electronic medical records and statistically evaluating differences has proved successful in previous studies. Comparing patients in studies with the local clinic population from which they are drawn, rather than from national or international statistics, will support the implementation of representative recruitment.

Lessons learnt from such methods have enabled empowerment and facilitation of recruitment of underrepresented groups. For the GRACE trial this included community involvement, enrolment quotas and targeted public relations. The REPRIEVE study similarly co-developed recruitment best practices aided by structured interviews. Effective strategies including culturally sensitive information about clinical trials, practical assistance and peer support have been identified through similar research into the barriers to recruitment.

As a highly active well-established research unit co-located and strongly embedded within a large, diverse London clinic we are uniquely placed to put into practice lessons learned from this project. If successful, this study and project will provide tools to increase the diversity of the population in clinical trials in Harrison Wing to reach a position where the demographics of trial participants reflects that of the local population living with HIV. Direct benefits of this include increasing the generalizability of research results and increasing equality of access to what may be a patient's best treatment option. Importantly, Harrison Wing has a dynamic and established involvement in audit and Quality Improvement, enabling successful strategies to be implemented and improved upon sustainably.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for initial analysis to identify groups who are underrepresented:

* HIV positive
* ≥18 years old
* Registered to receive care under Harrison Wing (and thus potential candidates for Harrison Wing clinical studies) at any point in the period between 01/01/2017 and 31/12/2019 inclusive. The period 01/01/2017 and 31/12/2019 has been selected because it is recent, occurred prior to the disruption caused by the Covid-19 pandemic and there exists complete data regarding HIV clinical study participation during this time.

Inclusion criteria for Groups 1 and 2 of the virtual semi-structured interview aspect of this study:

Group 1:

* HIV positive
* ≥18 years old
* Currently registered to receive care under Harrison Wing (and thus potential candidates for Harrison Wing clinical studies)
* Has ≥ 1 demographic identified to be underrepresented as specified in 'trial statistics'
* Able and willing to provide written or witnessed informed consent to participate

Group 2:

* HIV positive
* ≥18 years old
* Currently registered to receive care under Harrison Wing
* Currently participating in any clinical study in which Harrison Wing is the/ a participating centre
* Able and willing to provide written or witnessed informed consent to participate

Inclusion criteria for self-administered surveys:

* HIV positive
* ≥18 years old
* Registered to receive care under Harrison Wing (and thus potential candidates for Harrison Wing clinical studies)

Exclusion Criteria:

-

Ages: 18 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: HIV Positive patients attend Harrison Wing Clinic, Guy's Hospital, London
Sampling Method: Non-Probability Sample
Enrollment: 3520 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Is being female associated with a lower chance of participating in the research study in Harrison Wing, Guy's Hospital, London | 12 months
  The primary outcome measure for the initial data analysis will be whether being female is associated with lower chance of taking part in a study within Harrison Wing, during the three year period 1st January 2017 to 31st December 2019.

CONTACTS AND LOCATIONS:
Overall Officials: Julianne Lwanga, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: Undecided